CLINICAL TRIAL: NCT04193982
Title: An Investigator Initiated Prospective, Four Arms Randomized Comparative Study of Efficacy and Safety of Saroglitazar, Vitamin E and Life Style Modification in Patients With Nonalcoholic Fatty Liver Disease (NAFLD)/ Non-alcoholic Steatohepatitis (NASH)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECR/346/Inst/AP/2013/RR-16
Record Dates: First submitted 2019-08-14; First posted 2019-12-11 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: NAFLD
Keywords: Saraglitazar; Vitamin E
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — saroglitazar; Vitamin E; Drug Combinations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Saraglitazar (Experimental): Patients will receive Saraglitazar 4 mg once daily for 6 months
  Interventions: Drug: Saroglitazar
- Vitamin E (Experimental): Patients will receive Vitamin E 400mg twice daily for 6 months
  Interventions: Drug: Vitamin E
- Combination (Experimental): Patients will receive combination of Saraglitazar 4 mg once daily and Vitamin E 400mg twice daily for 6 months
  Interventions: Drug: Combination drug
- Lifestyle (Active Comparator): Patients will follow instruction from dietician and life style changes advise as per protocol including targeting 7 to 10percent weight loss in 6 months
  Interventions: Behavioral: Lifestyle Changes

INTERVENTIONS:
Drug: Saroglitazar — Patient receives Saraglitazar 4mg once daily
  Arms: Saraglitazar
Drug: Vitamin E — Patient receive Vitamin E 400mg twice daily after food for 6 months
  Arms: Vitamin E
Drug: Combination drug — Patient receives Vitamine E 400mg twice daily and Saraglitazar 4 mg once daily for 6 months
  Arms: Combination
Behavioral: Lifestyle Changes — Patients receives dietary advise and does exercise in form of aerobic and targets 7 to 10 percent weight loss in 6 months
  Arms: Lifestyle

SUMMARY:
Saroglitazar and Vitamin E are both being extensively used in India for non alcoholic fatty liver disease, though none of these drugs are FDA approved for this indication.However they are backed up by number of studies which shows improvement in liver function , reduction in NAS score. However, there is no head to head trial , nor is there any study with a paired biopsy comparing two arms for a head to head study. We therefore designed this study to see the effect of Vitamin E vs Vitamin E plus saroglitazar vs Saroglitazar alone when compared to standard dietary and weight loss treatment for NAFLD with raised ALT levels.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adults (age 18 to 60) 2. Confirmed Diagnosis of NAFLD established either by imaging (ultrasound, CT scan or MRI) or liver biopsy showing simple steatosis, within 6 months of the Screening Phase for this study. The diagnosis of NAFLD is made according to the American Association for the Study of Liver Diseases (AASLD) criteria (Chalasaniet al.2017).

  1. There is hepatic steatosis by imaging or histology,
  2. There is no significant alcohol consumption,
  3. There are no competing etiologies for hepatic steatosis
  4. There are no co-existing causes for chronic liver disease. 3. Patient's demonstration of understanding of study requirements and treatment procedures, willingness to comply with all protocol-required evaluations.

     4. Either take biopsy proven NAFLD or imaging based NAFLD with ALT more than 1.5 times the upper limit of normal. (being considered as 32) 5. Liver biopsy would be done in selected cases where the cause of transaminitis was uncertain of possible biopsy would be done on case to case basis.

     Exclusion Criteria:
     1. Absence of regular or excessive use of alcohol within 2 years prior to initial screening. History of alcohol will be taken from the patient and one or more family member and patient will be defined as non-alcoholic if he/she is a total abstainer or takes >20g (males) or 10g (females) of alcohol per day or greater than 14 drinks per week in males or greater than 7 drinks per week in females. Approximately 10 g of alcohol equals one 'drink' unit. One unit equals 30 ml of distilled spirits, 355 ml beer, or 120 ml glass of wine.
     2. Presence of alternative causes of fatty liver, including:

        * Weight loss >10% in the 6 months before the Screening Visit
        * Total parenteral nutrition, starvation or protein-calorie malnutrition
        * Use of drugs associated with NAFLD for more than 12 consecutive weeks in the 1 year before start of the study, including amiodarone, tamoxifen, methotrexate, systemic glucocorticoids, anabolic steroids, tetracycline, estrogens in doses higher than used in oral contraceptives, vitamin A, L asparaginase, valproate, chloroquine, or antiretroviral drugs.
     3. History of bowel surgery, gastrointestinal (bariatric) surgery or undergoing evaluation for bariatric surgery for obesity, extensive small-bowel resection, or orthotopic liver transplants (OLT) or listed for OLT.
     4. History of other chronic liver disease (Viral hepatitis B or C, autoimmune hepatitis, cholestatic and metabolic liver diseases) and hemochromatosis.
     5. Patient has known cirrhosis (compensated /decompensated) either based on clinical criteria or liver histology or Imaging techniques.
     6. Patients with Hypothyroidism.
     7. Unstable cardiovascular disease, including:

        * unstable angina, (i.e., new or worsening symptoms of coronary heart disease within the past 3 months), acute coronary syndrome within the past 6 months, acute myocardial infarction in the past 3 months or heart failure of New York Heart Association class (III - IV) or worsening congestive heart failure, or coronary artery intervention, within the past 6 months
        * history of (within prior 3 months) or current unstable cardiac dysarrhythmias
        * uncontrolled hypertension (systolic BP>180 mmHg and/or diastolic BP >110 mmHg on two consecutive occasions)
        * stroke or transient ischemic attack within the prior 6 months
     8. History of myopathies or evidence of active muscle disease.
     9. History of malignancy in the past 5 years and/or active neoplasm with the exception of resolved superficial non-melanoma skin cancer.
     10. Participation in any other therapeutic clinical study in the past 3 months, including participation in any other NAFLD clinical trials.
     11. History of bladder disease and/or hematuria or has current hematuria except due to a urinary tract infection.
     12. Illicit substance abuse within the past 12 months.
     13. Pregnant/lactating female (including positive pregnancy test at the Screening Visit)
     14. History or other evidence of severe illness or any other conditions that would make the patient, in the opinion of the investigator, unsuitable for the study (such as poorly controlled psychiatric disease, HIV, coronary artery disease or active gastrointestinal conditions that might interfere with drug absorption).
     15. Patients who will not comply with diet and lifestyle changes can be excluded from the final analysis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-01-31 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Non alcoholic fatty liver fibrosis score at 8week, 16week and 24week. | 6 months
  Non alcoholic fatty liver fibrosis score would be assessed . This is a non invasive test calculated by the formula : -1.675 + 0.037 × age (years) + 0.094 × BMI (kg/m2) + 1.13 × IFG/diabetes (yes = 1, no = 0) + 0.99 × AST/ALT ratio - 0.013 × platelet (×109/l) - 0.66 × albumin (g/dl)
  Results are interpreted as :
  NAFLD Score < -1.455 = F0-F2 NAFLD Score -1.455 - 0.675 = indeterminate score NAFLD Score > 0.675 = F3-F4
  Change in the NAFLD fibrosis score from the initiation of treatment and at end of 6 months would be assessed.

SECONDARY OUTCOMES:
Serum Alanine aminotransferase (ALT) changes at 6 months. | 6 months
  Changes in Alanine aminotransferase at 6 months would be assessed.
Serum triglycerides (TG) level. | 6 months
  Improvement as evidenced by decrease in triglyceride at 6 months.
Change in fibrosis on Liver Biopsy at 6 months. | 6 months
  The study involves a paired liver biopsy and patients who undergo the second biopsy will be assessed for regression or decrease in fibrosis and steatosis score on biopsy.
  Score interpretation:
  Steatosis: < 5%- 0, 5-33%- 1, >33-66%- 2, >66%- 3. Fibrosis: F0- No fibrosis, F1- Mild fibrosis, F2- Moderate fibrosis, F3- Severe fibrosis
Serum Aspartate aminotransferase (AST) level at 6 months. | 6 months
  Changes in Aspartate aminotransferase at 6 months would be assessed.
Non alcoholic steatosis (NAS) score on liver biopsy at 6 months. | 6 months
  Change in Non alcoholic Steatosis (NAS) score at 6 months. NAS score interpretation: Range- 0 to 8
  ≥5- Non-alcoholic steatohepatitis (NASH)
Glycosylated Hemoglobin (HbA1C) Level at 6 months. | 6 months
  Change in glycosylated hemoglobin level (amount of glucose attached to hemoglobin) from baseline and at 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Asian Institute of Gastroenterology Hospitals, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Duseja A, Singh SP, Saraswat VA, Acharya SK, Chawla YK, Chowdhury S, Dhiman RK, Jayakumar RV, Madan K, Misra SP, Mishra H, Modi SK, Muruganathan A, Saboo B, Sahay R, Upadhyay R. Non-alcoholic Fatty Liver Disease and Metabolic Syndrome-Position Paper of the Indian National Association for the Study of the Liver, Endocrine Society of India, Indian College of Cardiology and Indian Society of Gastroenterology. J Clin Exp Hepatol. 2015 Mar;5(1):51-68. doi: 10.1016/j.jceh.2015.02.006. Epub 2015 Mar 6. PMID 25941433
- [Background] Dhiman RK, Duseja A, Chawla Y. Asians need different criteria for defining overweight and obesity. Arch Intern Med. 2005 May 9;165(9):1069-70. doi: 10.1001/archinte.165.9.1069-b. No abstract available. PMID 15883250
- [Background] Chalasani N, Younossi Z, Lavine JE, Diehl AM, Brunt EM, Cusi K, Charlton M, Sanyal AJ; American Gastroenterological Association; American Association for the Study of Liver Diseases; American College of Gastroenterologyh. The diagnosis and management of non-alcoholic fatty liver disease: practice guideline by the American Gastroenterological Association, American Association for the Study of Liver Diseases, and American College of Gastroenterology. Gastroenterology. 2012 Jun;142(7):1592-609. doi: 10.1053/j.gastro.2012.04.001. Epub 2012 May 15. No abstract available. PMID 22656328
- [Background] Georgescu EF, Georgescu M. Therapeutic options in non-alcoholic steatohepatitis (NASH). Are all agents alike? Results of a preliminary study. J Gastrointestin Liver Dis. 2007 Mar;16(1):39-46. PMID 17410287
- [Background] Sanyal AJ, Brunt EM, Kleiner DE, Kowdley KV, Chalasani N, Lavine JE, Ratziu V, McCullough A. Endpoints and clinical trial design for nonalcoholic steatohepatitis. Hepatology. 2011 Jul;54(1):344-53. doi: 10.1002/hep.24376. PMID 21520200